CLINICAL TRIAL: NCT05144646
Title: Peripheral Tissue Perfusion and Oxygenation in Areas at Risk of Deterioration of Skin Integrity Subjected to Treatment With Hyperoxygenated Fatty Acids vs Virgin Olive Oil
Brief Title: Peripheral Tissue Perfusion and Oxygenation in Areas at Risk of Press Ulcer (POTER-OIL)
Acronym: POTER-OIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: JOSE MIGUEL MORALES ASENCIO (Other)
Responsible Party: Sponsor-Investigator, JOSE MIGUEL MORALES ASENCIO, University Professor Vice Dean of Research and Postgraduate Studies Coordinator of the Doctoral Program in Health Sciences Faculty of Health Sciences., University of Malaga
Organization: University of Malaga (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI21/01197
Record Dates: First submitted 2021-11-07; First posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Pressure Ulcer
Keywords: Hyperoxygenated fatty acid; Olive oil; Prevention; Perfusion and Oxygenation
MeSH Terms: conditions — Pressure Ulcer | interventions — Mepentol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEALTHY SUBJECTS (Experimental): With healthy subjects in a randomised, open experimental design, in an intrasubject control group (application of HFA / EVOO on one heel, using the contralateral heel as a control and evaluating oxygenation and tissue perfusion in both cases). This intervention would correspond to phase 1
  Interventions: Other: MEPENTOL® AND FARMAOLIVA® IN HEALTHY WITH INTRASUBJECT CONTROL
- PATIENTS (Experimental): With hospitalised patients and patients from social and health centers an experimental, randomised, open design, also with an intrasubject control group (application of HFA / EVOO on one heel, using the contralateral heel as a control and evaluating oxygenation and tissue perfusion in both cases). This intervention would correspond to phase 2.
  Interventions: Other: MEPENTOL® AND FARMAOLIVA® IN PATIENTS WITH INTRASUBJECT CONTROL

INTERVENTIONS:
Other: MEPENTOL® AND FARMAOLIVA® IN HEALTHY WITH INTRASUBJECT CONTROL — The corresponding product (HFA -Mepentol®- or EVOO - Farmaoliva®- depending on the study group assigned) will be applied to the subject's right heel, while the contralateral, left, heel will remain as a control. To ensure that the product is completely absorbed into the skin, the subject will then be asked to remain lying face up, at an angle of 30º to the bed, for one hour. The Doppler and infrared laser probes will then be placed on each heel (on the calcaneal tuberosity), for approximately four hours. The subjects will be asked to keep their lower body immobile, but will be able to move their arms and neck gently. Average values for capillary blood flow, local temperature and tissue oxygenation will be collected at 15-minute intervals, although the first 15-minute reading, while the parameters are becoming established, will be discarded.
  Arms: HEALTHY SUBJECTS
Other: MEPENTOL® AND FARMAOLIVA® IN PATIENTS WITH INTRASUBJECT CONTROL — In the second, clinical phase, the measurement protocol will be different, although certain aspects will remain unchanged. The product in question (HFA -Mepentol®- or EVOO -Farmaoliva®- according to the randomisation group assigned) will be applied to the intervention heel (right), leaving the contralateral (left) heel as a control. In addition, every patient will receive the standard PU prevention measures described in the protocol applicable for persons at risk of this condition. The intervention will be carried out in the morning, after bathing, as is customary in acute-care hospital units. The data will be collected at 15-minute intervals, although the first interval will be discarded, as described above. This procedure will be repeated every day during hospitalisation, to assess the cumulative action of the barrier cream. Each measurement will last approximately one hour each day.
  Arms: PATIENTS

SUMMARY:
The study objectives will be:

Primary objectives:

1. To determine the effects on oxygenation and tissue perfusion of applying HFA (Hyperoxygenated Fatty Acids) or EVOO (Extra Virgin Olive Oil) to the heels of healthy subjects, evaluating the maximum variation of oxygenation and flow when the heels are subjected to pressure.
2. To determine the levels of tissue oxygenation and perfusion associated with the appearance of blanching erythema in the heels of acute hospitalised patients and patients admitted to social health centers for the elderly.

Secondary objectives:

1. To determine whether there are differences in oxygenation and peripheral tissue perfusion between heels to which HFA vs. EVOO is applied.
2. To evaluate the possible progressive loss of the efficacy of HFA and EVOO in terms of tissue oxygenation and perfusion in patients who are bedridden for extended periods.

Methodology:

Experimental study in two phases: preclinical and clinical. Phase 1 with healthy subjects, with a randomized and open design, with an intrasubject control group. Phase 2 with hospitalized subjects and patients admitted to social health centers for the elderly, with a randomized and open design, with an intrasubject control group.

DETAILED DESCRIPTION:
The study participants will be subjected to simple randomisation to receive HFA or EVOO . The phase 1 will be carried out in healthy volunteers recruited at the Faculty of Health Sciences in the University of Malaga (Spain). Inclusion criteria: Healthy volunteers, aged >20 years, with no cardiovascular, neurological, digestive, endocrine, renal, gynaecological, respiratory, haematological, infectious, dermatological, autoimmune or osteomuscular diseases diagnosed, nor functional limitations, with objective tissue integrity, BMI of 18.5-25.9 kg/cm2 and no scars on the heels.

The phase 2 will be carried out patients admitted to acute hospitalised patients and patients admitted to social health centers for the elderly, at risk of deterioration of skin integrity according to Braden score <16, no presence of PU, who agree to participate in the study.

Measurement instruments Perfusion and tissue temperature data will be obtained by laser doppler flowmetry (LDF), with MoorVMS-LDF equipment. This system has two monitoring probes (one for each heel) that are brought into contact with the skin. The laser light is transmitted through an optical fibre to the tissue, reaching a depth of approximately 1 mm. The scattered light is collected by optical fibres and, at the same time, transmitted to a photodetector. The system has a measuring range of 5-50º C, a resolution of 0.1º C and an accuracy of ± 0.3º C.

Tissue oxygenation will be measured by near-infrared spectroscopy, with the MoorVMS-NIRS instrument. As in the previous case, the system contains two monitoring probes that are placed in contact with the skin. This method measures oxygen saturation (SpO2), which is calculated from absolute concentrations of oxygenated and deoxygenated haemoglobin in the tissue. Each probe consists of a detector head, containing two identical photodiodes, and an emitter head, with two infrared LEDs that emit light at approximately 750-850 nm. The system has a measurement range of 0-99%, a resolution of 1% and an accuracy of ± 3%.

All information on capillary blood flow, local temperature and tissue oxygenation will be monitored continuously and simultaneously using appropriate software. All measurement procedures are non-invasive. Both Moor instruments are certified to ISO 13485: 2016.

ELIGIBILITY:
PHASE ONE HEALTHY SUBJECTS

Inclusion criteria:

* Healthy volunteers, aged > 20 years without functional limitation.
* BMI of 18.5-25.9 kg/cm2.
* No scars on the heels.

Exclusion criteria:

* Failure to meet all of the above criteria.
* Smokers.
* Consume high levels of alcohol (> 20g/week).
* Tattoos in the measurement areas.

PHASE TWO - PATIENTS

Inclusion criteria:

* Patients aged > 20.
* Patients with risk of deterioration of skin integrity according to Braden score <16.
* no presence of Press Ulcer.

Exclusion criteria:

* Presence of vasoactive drugs in infusion
* Subjects with a pacemaker and/or implanted defibrillator.
* Fever and anaemia with Hb <10 g/dl.
* Hypotension with systolic blood pressure <80 mmHg.
* Transfusion during the last four weeks.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2022-01-04 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Perfusion and tissue temperature | In the healthy group, measurements will be made for four hours at fifteen-minute intervals for 1 day. In the hospitalized patients group, measurements will be made for one hour at fifteen-minute intervals every day for 7 days.
  Perfusion and tissue temperature data will be obtained by laser doppler flowmetry (LDF), with MoorVMS-LDF equipment. This system has two monitoring probes (one for each heel) that are brought into contact with the skin. The laser light is transmitted through an optical fibre to the tissue, reaching a depth of approximately 1 mm. The scattered light is collected by optical fibres and, at the same time, transmitted to a photodetector. The system has a measuring range of 5-50º C, a resolution of 0.1º C and an accuracy of ± 0.3º C.
Tissue oxygenation | In the healthy group, measurements will be made for four hours at fifteen-minute intervals for 1 day. In the hospitalized patients group, measurements will be made for one hour at fifteen-minute intervals every day for 7 days.
  Tissue oxygenation will be measured by near-infrared spectroscopy, with the MoorVMS-NIRS instrument. As in the previous case, the system contains two monitoring probes that are placed in contact with the skin. This method measures oxygen saturation (SpO2), which is calculated from absolute concentrations of oxygenated and deoxygenated haemoglobin in the tissue. Each probe consists of a detector head, containing two identical photodiodes, and an emitter head, with two infrared LEDs that emit light at approximately 750-850 nm. The system has a measurement range of 0-99%, a resolution of 1% and an accuracy of ± 3%.

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Lupiáñez Pérez, PhD, Principal Investigator — Faculty of Health Sciences, University of Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avsar P, Moore Z, Patton D, O'Connor T, Budri AM, Nugent L. Repositioning for preventing pressure ulcers: a systematic review and meta-analysis. J Wound Care. 2020 Sep 2;29(9):496-508. doi: 10.12968/jowc.2020.29.9.496. PMID 32924821
- [Background] Bail K, Draper B, Berry H, Karmel R, Goss J. Predicting excess cost for older inpatients with clinical complexity: A retrospective cohort study examining cognition, comorbidities and complications. PLoS One. 2018 Feb 23;13(2):e0193319. doi: 10.1371/journal.pone.0193319. eCollection 2018. PMID 29474407
- [Background] Coleman S, Gorecki C, Nelson EA, Closs SJ, Defloor T, Halfens R, Farrin A, Brown J, Schoonhoven L, Nixon J. Patient risk factors for pressure ulcer development: systematic review. Int J Nurs Stud. 2013 Jul;50(7):974-1003. doi: 10.1016/j.ijnurstu.2012.11.019. Epub 2013 Feb 1. PMID 23375662
- [Background] Diaz-Valenzuela A, Garcia-Fernandez FP, Carmona Fernandez P, Valle Canete MJ, Pancorbo-Hidalgo PL. Effectiveness and safety of olive oil preparation for topical use in pressure ulcer prevention: Multicentre, controlled, randomised, and double-blinded clinical trial. Int Wound J. 2019 Dec;16(6):1314-1322. doi: 10.1111/iwj.13191. Epub 2019 Sep 2. PMID 31475465
- [Background] Ferris A, Price A, Harding K. Pressure ulcers in patients receiving palliative care: A systematic review. Palliat Med. 2019 Jul;33(7):770-782. doi: 10.1177/0269216319846023. Epub 2019 Apr 24. PMID 31018829
- [Background] Gallart, E., Fuentelsaz, C., Vivas, G., Garnacho, I., Font, L., & Arán, R. (2001). Estudio experimental para comprobar la efectividad de los ácidos grasos hiperoxigenados en la prevención de las úlceras por presión en pacientes ingresados. Enfermería Clínica, 11(5), 179-183. https://doi.org/10.1016/s1130-8621(01)73714-x
- [Background] Gaspar S, Peralta M, Marques A, Budri A, Gaspar de Matos M. Effectiveness on hospital-acquired pressure ulcers prevention: a systematic review. Int Wound J. 2019 Oct;16(5):1087-1102. doi: 10.1111/iwj.13147. Epub 2019 Jul 1. PMID 31264345
- [Background] Gomez-Gonzalez AJ, Morilla-Herrera JC, Lupianez-Perez I, Morales-Asencio JM, Garcia-Mayor S, Leon-Campos A, Marfil-Gomez R, Aranda-Gallardo M, Moya-Suarez AB, Kaknani-Uttumchandani S. Perfusion, tissue oxygenation and peripheral temperature in the skin of heels of healthy participants exposed to pressure: a quasi-experimental study. J Adv Nurs. 2020 Feb;76(2):654-663. doi: 10.1111/jan.14250. Epub 2019 Nov 20. PMID 31651050
- [Background] Jull A, McCall E, Chappell M, Tobin S. Measuring hospital-acquired pressure injuries: A surveillance programme for monitoring performance improvement and estimating annual prevalence. Int J Nurs Stud. 2016 Jun;58:71-79. doi: 10.1016/j.ijnurstu.2016.02.005. Epub 2016 Feb 17. PMID 27087299
- [Background] Lazaro-Martinez JL, Lopez-Moral M, Garcia-Alamino JM, Bohbot S, Sanz-Corbalan I, Garcia-Alvarez Y. Evolution of the TcPO2 values following hyperoxygenated fatty acids emulsion application in patients with diabetic foot disease: results of a clinical trial. J Wound Care. 2021 Jan 2;30(1):74-79. doi: 10.12968/jowc.2021.30.1.74. PMID 33439078
- [Background] Lechner A, Kottner J, Coleman S, Muir D, Beeckman D, Chaboyer W, Cuddigan J, Moore Z, Rutherford C, Schmitt J, Nixon J, Balzer K. Outcomes for Pressure Ulcer Trials (OUTPUTs) project: review and classification of outcomes reported in pressure ulcer prevention research. Br J Dermatol. 2021 Apr;184(4):617-626. doi: 10.1111/bjd.19304. Epub 2020 Jul 27. PMID 32510579
- [Background] Li Z, Lin F, Thalib L, Chaboyer W. Global prevalence and incidence of pressure injuries in hospitalised adult patients: A systematic review and meta-analysis. Int J Nurs Stud. 2020 May;105:103546. doi: 10.1016/j.ijnurstu.2020.103546. Epub 2020 Jan 31. PMID 32113142
- [Background] Lindgren M, Malmqvist LA, Sjoberg F, Ek AC. Altered skin blood perfusion in areas with non blanchable erythema: an explorative study. Int Wound J. 2006 Sep;3(3):215-23. doi: 10.1111/j.1742-481X.2006.00238.x. PMID 16984577
- [Background] Lovegrove J, Fulbrook P, Miles SJ, Steele M. Effectiveness of interventions to prevent pressure injury in adults admitted to acute hospital settings: A systematic review and meta-analysis of randomised controlled trials. Int J Nurs Stud. 2021 Oct;122:104027. doi: 10.1016/j.ijnurstu.2021.104027. Epub 2021 Jun 30. PMID 34334175
- [Background] Lovegrove J, Fulbrook P, Miles S, Steele M. Effectiveness of interventions to prevent pressure injury in adults admitted to intensive care settings: A systematic review and meta-analysis of randomised controlled trials. Aust Crit Care. 2022 Mar;35(2):186-203. doi: 10.1016/j.aucc.2021.04.007. Epub 2021 Jun 16. PMID 34144865
- [Background] Lupianez-Perez I, Morilla-Herrera JC, Kaknani-Uttumchandani S, Lupianez-Perez Y, Cuevas-Fernandez-Gallego M, Martin-Santos F, Caro-Bautista J, Morales-Asencio JM. A cost minimization analysis of olive oil vs. hyperoxygenated fatty acid treatment for the prevention of pressure ulcers in primary healthcare: A randomized controlled trial. Wound Repair Regen. 2017 Sep;25(5):846-851. doi: 10.1111/wrr.12586. Epub 2017 Nov 6. PMID 28922519
- [Background] Lupianez-Perez I, Uttumchandani SK, Morilla-Herrera JC, Martin-Santos FJ, Fernandez-Gallego MC, Navarro-Moya FJ, Lupianez-Perez Y, Contreras-Fernandez E, Morales-Asencio JM. Topical olive oil is not inferior to hyperoxygenated fatty aids to prevent pressure ulcers in high-risk immobilised patients in home care. Results of a multicentre randomised triple-blind controlled non-inferiority trial. PLoS One. 2015 Apr 17;10(4):e0122238. doi: 10.1371/journal.pone.0122238. eCollection 2015. PMID 25886152
- [Background] Maki-Turja-Rostedt S, Stolt M, Leino-Kilpi H, Haavisto E. Preventive interventions for pressure ulcers in long-term older people care facilities: A systematic review. J Clin Nurs. 2019 Jul;28(13-14):2420-2442. doi: 10.1111/jocn.14767. Epub 2019 Jan 25. PMID 30589987
- [Background] Pancorbo Hidalgo, P. L., García Fernández, F. P., Pérez López, C., & Soldevilla Agreda, J. J. (2019). Prevalencia de lesiones por presión y otras lesiones cutáneas relacionadas con la dependencia en población adulta en hospitales españoles: resultados del 5o Estudio Nacional de 2017. Gerokomos, 30(2), 76-86. http://www.scielo.org.co/scielo.php?script=sci_arttext&pid=S2011-08392020000400014&lang=es%0Ahttp://www.scielo.org.co/pdf/unmed/v61n4/2011-0839-unmed-61-04-00014.pdf
- [Background] Pittman J, Beeson T, Dillon J, Yang Z, Cuddigan J. Hospital-Acquired Pressure Injuries in Critical and Progressive Care: Avoidable Versus Unavoidable. Am J Crit Care. 2019 Sep;28(5):338-350. doi: 10.4037/ajcc2019264. PMID 31474603
- [Background] Shi C, Dumville JC, Cullum N. Skin status for predicting pressure ulcer development: A systematic review and meta-analyses. Int J Nurs Stud. 2018 Nov;87:14-25. doi: 10.1016/j.ijnurstu.2018.07.003. Epub 2018 Jul 8. PMID 30015089
- [Background] Tisserand G, Zenati N, Seinturier C, Blaise S, Pernod G. Prevalence and severity of peripheral arterial disease among patient with heel pressure ulcer: a retrospective study of 42 patients. Geriatr Psychol Neuropsychiatr Vieil. 2017 Sep 1;15(3):242-246. doi: 10.1684/pnv.2017.0680. PMID 28872035
- [Background] Torra-Bou, J. E., Pérez-Acevedo, G., Bosch-Alcaraz, A., García-Fernández, F. P., Sarabia-Lavin, R., Soldevilla-Agreda, J. J., & Verdú-Soriano, J. (2020). Pressure injury incidence in pediatric and neonatal intensive care units: Systematic review (2000-2016). Gerokomos, 31(3), 180-192. https://doi.org/10.4321/S1134-928X2020000300010
- [Background] Torra-Bou, J.-E., García-Fernández, F.-P., Pérez-Acevedo, G., Sarabia-Lavin, R., Paras-Bravo, P., Rodríguez-Palma, M., & Verdú-Soriano, J. (2017). El impacto económico de las lesiones por presión. Revisión bibliográfica integrativa. Gerokomos (Madr., Ed. Impr.), 28(2), 83-87. https://scielo.isciii.es/scielo.php?script=sci_arttext&pid=S1134-928X2017000200083
- [Background] VanGilder C, Lachenbruch C, Algrim-Boyle C, Meyer S. The International Pressure Ulcer Prevalence Survey: 2006-2015: A 10-Year Pressure Injury Prevalence and Demographic Trend Analysis by Care Setting. J Wound Ostomy Continence Nurs. 2017 Jan/Feb;44(1):20-28. doi: 10.1097/WON.0000000000000292. PMID 27977509